CLINICAL TRIAL: NCT04177654
Title: Establishing a Surveillance System to Monitor the Global Patterns of Drug Efficacy and Emergence of Anthelmintic Resistance in Soil-transmitted Helminth Programs
Brief Title: Monitoring Drug Efficacy and Anthelmintic Resistance in Soil-transmitted Helminth Programs
Acronym: StarwormsWP2
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: OPP1120972_WP2
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Soil-transmitted Helminth Infections
Keywords: parasitology; helminth infections; Ascaris; Trichuris; hookworm; qPCR; microscopy; drug resistance; diagnosis; drug efficacy
MeSH Terms: conditions — Trematode Infections; Ancylostomiasis; Disease | interventions — Benzimidazoles; Albendazole; Mebendazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool samples preserved in Ethanol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Cambodia: The group of school-aged children from Cambodia who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Bangladesh: The group of school-aged children from Cambodia who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Vietnam: The group of school-aged children from Vietnam who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Lao PDR: The group of school-aged children from Lao PDR who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Ghana: The group of school-aged children from Ghana who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Senegal: The group of school-aged children from Senegal who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Rwanda: The group of school-aged children from Rwanda who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles
- Haiti: The group of school-aged children from Haiti who are being screened. Children will receive a single standard dose of benzimidazole drug (either 400mg of Albendazole or 500mg of Mebendazole) and stool samples will be collected prior to and 2-3 weeks following treatment.
  Interventions: Drug: Benzimidazoles

INTERVENTIONS:
Drug: Benzimidazoles — A single dose of benzimidazole drug (400mg Albendazole or 500mg Mebendazole) will be administered as part of routine deworming services.
  Other Names: Albendazole; Mebendazole

SUMMARY:
Soil-transmitted helminths (STHs) are a group of parasitic worms that infect millions of children in sub-tropical and tropical countries, resulting in malnutrition, growth stunting, intellectual retardation and cognitive deficits. To control the morbidity due to these worms, school-based deworming programs are implemented, in which anthelminthic drugs are administered to children without prior diagnosis. The continued fight against these worms is aided by the London declaration on neglected tropical diseases, which helps sustain and expand global drug donation program, resulting in an unprecedented growth of deworming programs. However, the high degree of drug pressure makes deworming programs vulnerable to the development of anthelmintic resistance because they only rely on one drug with sometimes suboptimal efficacy and there is no availability of alternative drugs. Moreover, at present, there is no surveillance system to monitor the emergence and spread of anthelmintic resistance. It remains unclear to what extent the efficacy of drugs may have dropped and whether anthelmintic resistance is already present. This project aims to strengthen the monitoring and surveillance of drug efficacy and anthelmintic resistance in STH programs. As such, it will support deworming programs in their quest to eliminate STHs as a public health problem. The overall aim of this study is to pilot a surveillance system to assess anthelmintic drug efficacy and the emergence of AR in 9 countries were drug pressure has been high over a long period of time.

The specific objectives are to:

1. Assess the prevalence of moderate/heavy intensity infections of the different STH
2. Assess the drug efficacy of a single dose of BZ drugs against STH infections in these countries
3. Assess the frequency of the ß-tubulin SNPs linked to BZ resistance
4. Identify implementation-related barriers and opportunities for monitoring drug efficacy and AR in national PC programs for STH.
5. Expand the Starworms repository of STH field samples

DETAILED DESCRIPTION:
Soil-transmitted helminths (STHs) include Ascaris lumbricoides, Trichuris trichiura, and two hookworm species, namely Necator americanus and Ancylostoma duodenale. They are responsible for the highest burden among all neglected tropical diseases (NTDs). Recent global estimates indicate that in 2010 more than 1.4 billion people were infected with at least one of the four STH species, resulting in a global burden of approximately 3.3 million disability-adjusted life years (DALYs). To control the morbidity caused by STHs, preventive chemotherapy (PC) is the main strategy. This entails the periodical administration of a single-oral dose of albendazole (ALB; 400 mg) or mebendazole (MEB; 500 mg) to at-risk populations (ie., preschool-aged (preSAC), school-aged children (SAC) and women of reproductive age) (WHO, 2017). Accelerated by the London Declaration on NTDs, the global coverage of children in PC programs has increased from ~30% in 2011 to 63.6% in 2016, with the goal of covering at least 75% of children by 2020. The laudable long-term aim is to eliminate STHs as a public health problem (<1% moderate/heavy intensity infections), and to eventually declare targeted geographical areas free of infections.

This high level of drug pressure makes PC programs highly vulnerable to the development of anthelmintic resistance (AR). First, the community relies on two drugs (ALB and MEB) of the same class (benzimidazole (BZ) drugs), and with the same mode of action (the inhibition of the polymerization of microtubules). Hence the emergence of AR is likely to occur as drug donations expand. This has been substantiated in veterinary medicine, where AR has developed within a decade of the introduction of every anthelmintic class. Moreover, the development of AR against one BZ drug would most likely be accompanied by poor anthelmintic drug efficacy of the other BZ drug. Second, drugs are administered in single doses. Although a single dose is operationally justified, it never achieves 100% efficacy. Consequently, this practice may further select for the development of AR when suboptimal doses are widely applied over a significant period. Finally, only few anthelmintic drugs are licensed for the treatment of STH infections in humans Thus, should AR against BZ drugs eventually emerge and spread, PC-based control of STHs will be even more limited than at present with few acceptable alternative options. Hence, this re-enforces the urgent necessity for increased accessibility of anthelmintic drugs of different anthelmintic classes and thoroughly designed surveillance systems that allow detection of any changes in anthelmintic drug efficacy arising through the evolution of AR in these helminths.

Currently, any global surveillance system to monitor both drug efficacy and emergence of AR is lacking, and as a consequence it remains unclear to what extent the efficacy of drugs may have dropped and whether AR is already present. One of the main reasons for this lack of monitoring systems is the absence of a framework that guides and supports healthcare decision makers in planning, performing and reporting surveys. The development of such a framework is not straightforward. Moreover, PC programs typically operate in resource-limitedsettings, and therefore it is indispensable that health-care decision makers have some pliancy to minimize both financial and technical resources, while assuring a reliable assessment of the drug efficacy and spread of AR.

To conclude, AR is a real threat for PC programs targeting human STHs. To establish a surveillance system, and to hence further ensure the efficacy of the administered drugs, there is a need for diagnostic methods that effectively mitigate important obstacles of performing, analysing and reporting drug efficacy surveys in resource poor settings, and a validated molecular marker to detect emergence of AR at an early stage. Subsequently, a surveillance system should be established to assess global patterns of drug efficacy and AR. Finally, tools for planning routine AR monitoring, and for following up the global changes in drug efficacy and spread of AR over time should be made available.

The overall aim of this study is to pilot a surveillance system to assess anthelmintic drug efficacy and the emergence of AR in 11 countries were PC coverage has been high over a long period of time. The specific objectives are to:

1. Assess the prevalence of moderate/heavy intensity infections of the different STH
2. Assess the drug efficacy of a single dose of BZ drugs against STH infections in these countries
3. Assess the frequency of the ß-tubulin SNPs linked to BZ resistance
4. Measure the costs related to monitoring drug efficacy and AR in national PC programs for STH.
5. Expand the Starworms repository of STH field samples

A series of drug efficacy trials will be performed in 9 STH endemic countries (Lao PDR, Bangladesh, Vietnam, Cambodia, Senegal, Ghana, Rwanda, Haiti) during their national PC program. These trials were designed to correctly classify the efficacy of a single oral dose of BZ drugs against STH infections in SAC into 'normal', 'doubtful' and 'reduced'. The study will focus on SAC (age 5-14) since they are the major target population of PC programs against STH, and they usually represent the group with highest intensity of infection for A. lumbricoides and T. trichiura. At baseline, SAC will be asked to provide a fresh stool sample. All children that meet all inclusion criteria and none of the exclusion criteriawill be enrolled in the study. They will be treated with a single oral dose of BZ drug under supervision. The choice of BZ drug will depend on the drug used in the STH program. The drug used in the study will be provided by the national PC program.

All collected stool samples at baseline will be processed to determine the fecal egg counts (FECs; expressed in eggs per gram of stool (EPG)) for each STH using a duplicate Kato-Katz thick smear. Positive baseline samples will be preserved for further molecular analysis. Fourteen to 21 days after drug administration, a second stool sample will be collected from all the children that were excreting eggs of any STH at baseline. These stool samples will again be examined by a duplicate Kato-Katz thick smear. All follow-up samples will be preserved for further molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, is 5-14 years of age
* Subject is otherwise in healthy condition (based on medical history and physical examination)
* Parent(s)/guardians of subject signed an informed consent document indicating that they understand the purpose of and procedures required for the study and that they are willing to have their child participate in the study
* Subject of ≥6 years has assented to participate in the study
* Subject of ≥12 years has signed an informed consent document indicating that they understand the purpose of the study and procedures required for the study and are willing to participate in the study
* Subject has provided a stool sample of at least 5 grams.

Exclusion Criteria:

* Subject has active diarrhoea (defined as the passage of 3 or more loose or liquid stools per day) at baseline or follow-up.
* Subject has an acute medical condition or is experiencing a severe concurrent medical condition
* Subject has a known hypersensitivity to ALB or MEB
* Subject has received anthelmintic treatment within 90 days prior to the start of the treatment
* Subject vomited within 4 hours following drug ingestion.
* Subject is not able to provide a stool sample of minimum 5 grams at baseline or follow-up.
* Subject has not swallowed the entire tablet.

Ages: 5 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Healthy school-aged children aged 5-14.
Sampling Method: Non-Probability Sample
Enrollment: 9457 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
moderate/heavy intensity infections of the different STH | up to 12 months
  The data collected at baseline (prior to treatment) will provide valuable information on the infection intensities and prevalence of the different STH in that population.
drug efficacy of a single dose of BZ drugs against STH infections in these countries | up to 12 months
  The reduction in egg output of the cohort of infected school aged children will inform us on the efficacy of the administered drug.
frequency of the ß-tubulin SNPs linked to BZ resistance | up to 12 months
  The collected stool samples will be analyzed and SNPs linked to benzimidazole drug resistance in STH will be quantified using molucular techniques like pyrosequencing, whole gene sequencing and LAMP.

SECONDARY OUTCOMES:
costs related to monitoring drug efficacy and AR in national PC programs for STH. | up to 12 months
  The absolute cost of the different drug efficacy studies will be evaluated using a standardized cost-description protocol to help provide a general estimate of the cost of implementing routine drug efficacy studies in endemic areas.
Expand the Starworms repository of STH field samples | up to 12 months
  The collection of stool samples will provide a valuable addition to the Starworms repository of STH field samples which can serve other research.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Levecke, PhD, Principal Investigator — University Ghent
Locations (8):
- Filariasis Elimination, STH Control and Little Doctor Program, Communicable Disease Control (CDC),Directorate General of Health Services (DGHS), MOHFW, Dhaka, Bangladesh
- Ministry of Health, Cambodia, Phnom Penh, Cambodia
- Centre for Science and Industrial Research, Accra, Ghana
- PAHO, Port-au-Prince, Haiti
- Centre for Malariology, Parasitology and Entomology Lao PDR, Vientiane, Laos
- Rwanda Biomedical Center/Ministry of Health of Rwanda - NTD&OPD Unit, Kigali, Rwanda
- NTD Programme, Ministry of Health, Dakar, Senegal
- Institute of Malariology Parasitology and Entomology (Nimpe),, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified results will be shared online and with collaborating researchers for further extensive analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No specific time-frame will be applied.
Access Criteria: Free access for all
URL: https://www.starworms.org/tools/overview/starworms-documents

REFERENCES:
- See also: Project homepage — http://www.starworms.org